CLINICAL TRIAL: NCT03416101
Title: Siewert Type II Esophageal Adenocarcinoma: on the Relationship Between Histology, Esophageal-gastric Intestinal Metaplasia and Gastric Greater Curvature Lymphatic Metastases, Survival
Brief Title: Siewert Type II Esophageal Adenocarcinoma: Relationship Between Histology and Survival
Acronym: SiewertIIEAC
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Sandro Mattioli, Associate Professor, University of Bologna
Other Study IDs: ADECC_2016
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Siewert Type II Adenocarcinoma of Esophagogastric Junction
Keywords: esophageal cancer; adenocarcinoma of the esophagus; esophageal surgery
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Surgical specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total Gastrectomy — The esophagus was resected at the arch level of the azygos vein, a frozen section of the resection margin was routinely performed to achieve a proximal clean resection margin. The surgical specimen was comprehensive of distal esophagus, stomach and omentum. Digestive tract continuity was established with Roux-en-Y esophagojejunostomy. Lymphadenectomy was extended to the thoracic stations R 2-4, 7-8-9, and L 4, numbered according to the Mountain's classification [39] (Suppl. File 2 Figure A) and to the abdominal stations 1-12, numbered according to the Japanese Research Society for Gastric Cancer (JRSGC) 1998 classification.
  Other Names: Distal Esophagectomy

SUMMARY:
In Siewert type II adenocarcinoma, the relationship between adenocarcinoma sub types and survival, histologic/biologic patterns related to the presence/absence of gastric greater curvature metastases, were investigated.

DETAILED DESCRIPTION:
In order to achieve further data on the biological patterns of intestinal and diffuse subtypes of esophageal adenocarcinoma (Lauren's classification), on the frequency of gastric greater curvature nodal stations and on the clinical relevance, in terms of prognosis and survival, of these parameters, a Siewert type II case series of Siewert type II adenocarcinomas, submitted to primary (no neoadjuvant therapy) surgical, studied, operated upon and followed up, were analysed. According to histologic patterns, cases were ordered in intestinal and diffuse adenocarcinoma sub types (Lauren's classification)and distinguished in Barret's, cardiopyloric, gastric types.

ELIGIBILITY:
Inclusion Criteria:

Siewert type II adenocarcinoma > 18 year submitted to primary surgery

Exclusion Criteria: Siewert type II adenocarcinoma submitted to neoadjuvant therapy.

Siewert type I adenocarcinoma. Siewert type III adenocarcinoma Squamous Carcinoma

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred fifty four Siewert type II cases were enrolled: 124 men (80.5%), 30 women (19.5%), median age 65.5 (interquartile range 58-71); Intestinal type 91 (59%) and Diffuse type 63 (41%).
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Survival | 5 years
  5 year survival between intestinal and diffuse types (Lauren's classification) of Siewert type II adenocarcinoma after primary surgery,

SECONDARY OUTCOMES:
Frequency of gastric greater curvature lymph nodes metastases in Siewert II adenocarcinoma | 5 years
  Frequency of gastric greater curvature lymph nodes metastases and survival

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Mattioli - Alma M Studiorum-University, MD, Principal Investigator — Department of Medical and Surgical Sciences
Locations (2):
- Italy (2):
  - Department of Medical and Surgical Sciences University of Bologna, Bologna, Bo
  - Sandro Mattioli - Alma Mater Studiorum-University, Bologna, BO

IPD SHARING:
Plan to Share IPD: No